CLINICAL TRIAL: NCT06228664
Title: Comparison of Bowen Therapy and Foam Rolling in Text Neck Syndrome Among Students
Brief Title: Bowen Therapy and Foam Rolling in Patients With Text Neck Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/MS-PT/01675 Kashmala Zeb
Record Dates: First submitted 2024-01-18; First posted 2024-01-29 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Neck Pain
Keywords: text neck syndrome; neck pain; bowen therapy; foam rolling
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- foam rolling (Active Comparator): foam rolling along with conventional physical therapy treatment
  Interventions: Other: foam rolling
- bowen therapy (Experimental): bowen therapy along with conventional physical therapy treatment
  Interventions: Other: bowen therapy

INTERVENTIONS:
Other: foam rolling — Foam Rolling Technique on trapezius and suboccipital muscles.conventional therapy (15 min Hot pack, neck isometric exercises and cervical ROM exercises within pain free range). Patients will be treated 3 times per week for 6 consecutive weeks
  Arms: foam rolling
Other: bowen therapy — Bowen Therapy. conventional therapy (15 min Hot pack, neck isometric exercises and cervical ROM exercises within pain free range) will be given to both groups. Patients will be treated 3 times per week for 6 consecutive weeks
  Arms: bowen therapy

SUMMARY:
This study aims to compare the effects of both the therapies on postural changes, pain, decreased ROM, and functional disability among students suffering from Text Neck Syndrome.

ELIGIBILITY:
Inclusion Criteria:

* neck-head trauma
* history of surgical intervention in the neck area
* neurological deficit
* severe neck pain which required medical treatment
* cervical disc disease with radiculopathy
* inflammatory or malignant type of pain
* systematic disease
* scoliosis
* kyphosis.

Exclusion Criteria:

* neck-head trauma
* history of surgical intervention in the neck area
* neurological deficit
* severe neck pain which required medical treatment
* cervical disc disease with radiculopathy
* inflammatory or malignant type of pain
* systematic disease
* scoliosis
* kyphosis.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-01-30 (Actual); Study Completion 2024-01-30 (Actual)

PRIMARY OUTCOMES:
Neck Disability Index | 6 week
  Changes from baseline, The neck disability index is a ten item self-reported questionnaire that assesses pain and associated disability, with a total max score of 50 points
NPRS | 6 week
  Changes from baseline.The Numeric Pain Rating Scale (NPRS) measures the subjective intensity of pain. The NPRS is an eleven-point scale from 0 to 10. "0" = no pain and "10" = most intense pain

CONTACTS AND LOCATIONS:
Overall Officials: Asmar Fatima, MS OMPT, Principal Investigator — Riphah International University
Locations (1):
- CECOS university of IT and emerging sciences, Peshawar, KPK, Pakistan

IPD SHARING:
Plan to Share IPD: No